CLINICAL TRIAL: NCT03370302
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-228 (a Catalytic TORC1/2 Inhibitor) as Single Agent in Adult East Asian Patients With Advanced Nonhematological Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) of TAK-228 as Single Agent in Adult East Asian Participants With Advanced Nonhematological Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: More favorable safety profile was observed in QD schedule, therefore further enrollment in QW schedule was terminated.
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C31008; U1111-1202-4296 (Registry Identifier: WHO); 1066064639 (Registry Identifier: Taiwan Ministry of Health and Welfare); 20170270241 (Other: Korea Food and Drug Administration); JapicCTI-183822 (Registry Identifier: Japan Ministry of Health)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2020-09-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Advanced Nonhematological Neoplasms
Keywords: Drug therapy
MeSH Terms: interventions — sapanisertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAK-228 Once Daily (Experimental): TAK-228, milled capsule, orally, once daily, on an empty stomach in a 28-day treatment cycle for up to 12 months or until disease progression or unacceptable toxicity or withdrawal of consent with a starting dose of 2 milligram (mg) in Cohort 1. Dose escalation will follow a standard 3+3 schema. If 2 mg, once daily, is safe and tolerable, then the dose will be escalated to 4 mg, once daily, until RP2D is determined.
  Interventions: Drug: TAK-228
- TAK-228 Once Weekly (Experimental): TAK-228, milled capsule, orally, once weekly, on an empty stomach in Cycle 1 of a 28-day treatment cycle and following a light meal from Cycle 2 for up to 12 months or until disease progression or unacceptable toxicity or withdrawal of consent with a starting dose of 20 mg in Cohort 1. Dose escalation will follow a standard 3+3 schema. If 20 mg, once weekly, is safe and tolerable, then the dose will be escalated to 30 mg, once weekly, until RP2D is determined.
  Interventions: Drug: TAK-228

INTERVENTIONS:
Drug: TAK-228 — TAK-228 Capsules.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, recommended phase 2 dose (RP2D), and to characterize PK of TAK-228 administered once daily or once weekly to East Asian participants with advanced nonhematological malignancies.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-228. TAK-228 is being tested to treat East Asian participants with advanced nonhematological malignancies for whom standard anticancer treatment is not available or is no longer effective. This study will assess the safety, tolerability, PK and will determine the RP2Ds of TAK-228.

The study will enroll approximately 46 participants, including at least 6 Japanese participants at RP2D dose level. Participants will be assigned to one of the following treatment arms:

* TAK-228 Once Daily
* TAK-228 Once Weekly

This multi-center trial will be conducted in South Korea, Taiwan, and Japan. The overall time to participate in this study is up to 12 months, unless in the opinion of the investigator and sponsor the participant would derive benefit from continued therapy beyond 12 months. Participants will be followed for 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. With advanced nonhematologic malignancies, with the exception of primary brain tumor, and have failed or are not eligible for standard of care therapy. History of brain metastasis may be allowed if all of the following criteria are met:

   * Brain metastases have been treated.
   * There is no evidence of progression or hemorrhage after treatment.
   * Steroid has been discontinued for >=4 weeks before the first dose of study drug.
   * There is no ongoing requirement for steroids or anti-epileptic drugs.
2. Received not more than 4 prior lines of systemic cytotoxic chemotherapy for advanced or metastatic disease.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
4. Screening clinical laboratory values as specified below:

   * Bone marrow reserve consistent with absolute neutrophil count (ANC) >=2000 per cubic millimeter (/mm^3), platelet count >=125,000/mm^3, and hemoglobin >=10 gram per deciliter (g/dL) without transfusion in the last 4 weeks.

Note: Prophylactic transfusions of blood products or any prophylactic use of hematopoietic growth factors (such as erythropoietin, thrombopoietin, granulocyte colony stimulating factor [G-CSF], and granulocyte macrophage colony stimulating factor [GM-CSF]) is not permitted during the screening period.

* Hepatic: Total bilirubin less than or equal to (<=) 1.5*upper limit of normal (ULN), alanine aminotransferase (ALT)/aspartate aminotransferase (AST) <=2.5*ULN (<=5*ULN if their elevation can be reasonably ascribed to the presence of hepatocellular carcinoma, biliary tract cancer, or metastatic disease in liver).
* Adequate renal function, defined as meeting any 1 of the following criteria:

  1. Serum creatinine <1.5*ULN.
  2. Creatinine clearance based on the Cockcroft-Gault estimate >=40 milliliter per minute (mL/min).
  3. Creatinine clearance based on urine collection (12- or 24-hour) >=40 mL/min.
  4. Metabolic: Glycosylated hemoglobin (hemoglobin A1c [HbA1c]) <=7%, fasting serum glucose <=130 milligram per deciliter (mg/dL), and fasting triglycerides <=300 mg/dL.

Exclusion Criteria:

1. Diagnosis of primary brain tumor.
2. Untreated brain metastasis or history of leptomeningeal disease or spinal cord compression.
3. Failed to recover from the reversible effects of prior anticancer therapies with the exception of alopecia, and after-effects associated with prior tyrosine kinase inhibitor therapy, such as hair depigmentation, hypothyroidism, and/or splinter hemorrhage.
4. Initiation of hematopoietic growth factors within 1 week before the first dose of study drug.
5. Manifestations of malabsorption caused by prior gastrointestinal surgery, gastrointestinal disease, or for some other reason that may alter the absorption of TAK-228. In addition, participants with enteric stomata are also excluded.
6. Poorly controlled diabetes mellitus defined as Hemoglobin A1c (HbA1c) greater than (>) 7%; participants with a history of transient glucose intolerance caused by corticosteroid administration are allowed if all other eligibility criteria are met.
7. Known human immunodeficiency virus infection.
8. Known hepatitis B surface antigen (HBsAg) positive, or known or suspected active hepatitis C virus (HCV) infection. Note: Participants who have isolated positive hepatitis B core antibody (HBcAb) and/or hepatitis B surface antibody (HBsAb) (that is, in the setting of negative HBsAg) may be enrolled but must have an undetectable hepatitis B virus (HBV) viral load. Participants who have positive hepatitis C virus antibody (HCVAb) may be enrolled but must have an undetectable HCV viral load.
9. Significant active cardiovascular or pulmonary disease before the first dose of study drug, including:

   * Uncontrolled hypertension (that is, systolic blood pressure >180 millimeter of mercury [mmHg]; diastolic blood pressure >95 mmHg).
   * Pulmonary hypertension.
   * Uncontrolled asthma or oxygen saturation less than (<) 90% by pulse oximetry on room air.
   * Significant valvular disease; severe regurgitation or stenosis by imaging independent of symptom control with medical intervention; or history of valve replacement.
   * Medically significant (symptomatic) bradycardia.
   * History of arrhythmia requiring an implantable cardiac defibrillator.
   * Baseline prolongation of the rate corrected QT interval (QTc) (example, repeated demonstration of QTc interval >480 millisecond [ms], or history of congenital long QT syndrome, or torsades de pointes).
10. Diagnosed or treated for another malignancy within 2 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chūōku, Tokyo-To
- Asan Medical Center, Seoul, South Korea
- National Taiwan-University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Shimizu T, Kuboki Y, Lin CC, Yonemori K, Yanai T, Faller DV, Dobler L, Gupta N, Sedarati F, Kim KP. A Phase 1 Study of Sapanisertib (TAK-228) in East Asian Patients with Advanced Nonhematological Malignancies. Target Oncol. 2022 Jan;17(1):15-24. doi: 10.1007/s11523-021-00855-w. Epub 2021 Nov 29. PMID 34843044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in Japan, South Korea and Taiwan from 17 January 2018 to 28 August 2019.
Pre-assignment Details: Participants with advanced nonhematological malignancies were enrolled in Dose Escalation and Expansion Phase to receive TAK-228 in 1 of the 2 schedules: once daily (QD) or once weekly (QW). Further enrollment in QW schedule was stopped and study was terminated before QW expansion because more favorable safety profile were observed in QD schedule.
Groups:
- Dose Escalation, Daily Dosing Arm: TAK-228 2 mg: TAK-228 2 milligram (mg), milled capsule, orally, once daily, on an empty stomach in a 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
- Dose Escalation, Daily Dosing Arm: TAK-228 3 mg: TAK-228 3 mg, milled capsule, orally, once daily, on an empty stomach in a 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
- Dose Escalation, Daily Dosing Arm: TAK-228 4 mg: TAK-228 4 mg, milled capsule, orally, once daily, on an empty stomach in a 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
- Dose Expansion, Daily Dosing Arm: TAK-228 3 mg: TAK-228 3 mg, milled capsule, orally, once daily, on an empty stomach in each 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
- Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg: TAK-228 20 mg, milled capsule, orally, once weekly, on an empty stomach in a 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
- Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg: TAK-228 30 mg milled, capsule, orally, once weekly, on an empty stomach in a 28-day treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
Period: Dose Escalation Phase
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Started | 3 | 6 | 7 | 0 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 7 | 0 | 3 | 3
Not completed — Other | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 4 | 2 | 0 | 3 | 1
Period: Dose Expansion Phase
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Started | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 6 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg | Total
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (5.20) | 55.8 (12.59) | 58.7 (10.36) | 56.3 (11.5) | 57.0 (6.93) | 54.0 (12.49) | 58 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 3 | 1 | 2 | 12
  Male | 2 | 4 | 4 | 3 | 2 | 1 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 7 | 6 | 3 | 3 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 4 | 3 | 3 | 3 | 1 | 17
  Taiwan, Province Of China | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Korea, Republic Of | 0 | 1 | 3 | 2 | 0 | 2 | 8
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 163.80 (10.000) | 167.05 (10.135) | 162.64 (5.839) | 162.42 (10.619) | 170.47 (12.003) | 160.73 (8.923) | 164.30 (8.96)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 63.33 (11.201) | 64.87 (13.958) | 62.09 (11.982) | 61.87 (17.490) | 61.43 (6.300) | 63.43 (10.001) | 62.84 (12.08)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 3 | 6 | 6 | 6 | 2 | 3 | 26
  Moderate Smoker (6-20 Cigarettes/ day) | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
Asian Sub-Category [Count of Participants; unit: Participants]
  Japanese | 3 | 4 | 3 | 3 | 3 | 1 | 17
  Korean | 0 | 1 | 3 | 2 | 0 | 2 | 8
  Chinese | 0 | 1 | 1 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug (up to Cycle 12 Day 58) (Cycle length= 28 days)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
Participants | 3 | 6 | 7 | 6 | 3 | 3

2. Primary Outcome: Number of Participants With Grade 3 or Higher TEAEs
Description: Adverse event (AE) Grades were evaluated as per National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE), version 4.03. Grade 1 scaled as Mild; Grade 2 scaled as Moderate; Grade 3 scaled as severe or medically significant but not immediately life-threatening; Grade 4 scaled as life-threatening consequences; and Grade 5 scaled as death related to AE.
Time Frame: Baseline up to 30 days after the last dose of study drug (up to Cycle 12 Day 58) (Cycle length= 28 days)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
Participants | 1 | 2 | 6 | 5 | 3 | 1

3. Primary Outcome: Number of Participants With Serious TEAEs
Time Frame: Baseline up to 30 days after the last dose of study drug (up to Cycle 12 Day 58) (Cycle length= 28 days)
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
Participants | 0 | 2 | 3 | 1 | 2 | 1

4. Primary Outcome: Dose Escalation Phase: Number of Participants With Dose-limiting Toxicities (DLTs) During Cycle 1
Description: Toxicity was evaluated according to NCI CTCAE version 4.03. DLT was defined as any of the following occurred events within the first 28 days of the administration of TAK-228 that were considered by investigator to be possibly related to therapy: Grade >=3 nonhematologic toxicity except for inadequately treated Grade 3 nausea and/or vomiting and diarrhea, Grade 3 hyperglycemia lasting <=14 days, Grade 3 rash lasting <=3 days; Grade 3 thrombocytopenia with hemorrhage or requiring platelet transfusion; Grade 3 anemia requiring blood transfusion; Grade 4 neutropenia lasting >7 days; Grade >=3 neutropenia of any duration with fever >=38.5 degree celsius and/or systemic infection; Any other >=Grade 4 hematologic toxicity; Inability to administer at least 75 percent (%) of planned doses of TAK-228 within Cycle 1 due to treatment-related toxicity and any clinically significant occurrence that the investigators and sponsor agreed would place participants at an undue safety risk.
Time Frame: Baseline up to Day 28 in Cycle 1 (Cycle length= 28 days)
Population: The DLT-evaluable set included participants who had received at least 75% of planned doses of TAK-228 in Cycle 1 unless interrupted by treatment-related events and had sufficient follow-up data considered by sponsor and investigator to determine whether DLT occurred.This outcome measure was planned to be assessed only in the dose escalation phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 3
Participants | 0 | 0 | 3 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Leading to Study Drug Discontinuation
Time Frame: Baseline up to 30 days after the last dose of study drug (up to Cycle 12 Day 58) (Cycle length= 28 days)
Population: The safety analysis set included all participants who received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
Participants | 1 | 0 | 2 | 0 | 0 | 1

6. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-228 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The pharmacokinetic (PK) analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
nanogram per milliliter (ng/mL) | 23.83 (9.6) | 41.35 (29.6) | 55.25 (26.2) | 41.78 (23.7) | 252.29 (75.2) | 268.61 (57.8)

7. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-228 on Cycle 1 Day 15
Time Frame: Cycle 1 Day 15 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The PK analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 3 | 3
ng/mL | 31.07 (48.6) | 46.85 (31.6) | 52.68 (47.2) | 45.02 (44.5) | 182.75 (70.5) | 364.58 (37.1)

8. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-228 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The PK analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
hours | 0.870 [0.50 to 2.03] | 0.990 [0.42 to 1.77] | 1.000 [0.50 to 2.00] | 0.500 [0.40 to 1.02] | 0.470 [0.40 to 2.08] | 1.970 [1.00 to 2.02]

9. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-228 on Cycle 1 Day 15
Time Frame: Cycle 1 Day 15 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 3 | 3
hours | 1.000 [0.50 to 2.08] | 0.965 [0.52 to 1.98] | 1.500 [0.92 to 3.00] | 1.000 [0.85 to 2.08] | 2.630 [1.97 to 4.10] | 2.000 [0.50 to 2.00]

10. Primary Outcome: Daily Dosing Arms, AUC24: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours for TAK-228 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: PK analysis set: Participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. This outcome measure was planned to be assessed only in Daily Dosing arms. Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 131.0311 (43.269) | 192.2467 (32.263) | 295.5497 (41.724) | 177.9464 (38.813)

11. Primary Outcome: Daily Dosing Arms, AUC24: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours for TAK-228 on Cycle 1 Day 15
Time Frame: Cycle 1 Day 15 pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg
Number analyzed (Participants) | 3 | 6 | 4 | 6
ng*hr/mL | 221.0132 (47.912) | 250.4458 (29.806) | 341.1219 (44.219) | 278.5369 (74.527)

12. Primary Outcome: Weekly Dosing Arms, AUC168: Area Under the Concentration-time Curve From 0 to 168 Hours for TAK-228 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length= 28 days)
Population: The PK analysis set included participants with sufficient dosing and PK data to reliably estimate 1 or more PK parameters. This outcome measure was planned to be assessed only in the Weekly Dosing arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 3
ng*hr/mL | 1636.7580 (49.907) | 2010.5661 (53.631)

13. Primary Outcome: Weekly Dosing Arms, AUC168: Area Under the Concentration-time Curve From 0 to 168 Hours for TAK-228 on Cycle 1 Day 15
Time Frame: Cycle 1 Day 15 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 3
ng*hr/mL | 1860.7705 (42.989) | 2958.0487 (47.602)

14. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From 0 to Time of Last Measurable Concentration for TAK-228 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
ng*hr/mL | 123.6468 (54.137) | 175.6252 (45.734) | 306.5602 (39.279) | 173.5642 (44.339) | 1471.9032 (45.692) | 1839.6167 (52.905)

15. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From 0 to Time of Last Measurable Concentration for TAK-228 on Cycle 1 Day 15
Time Frame: Cycle 1 Day 15 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 4 | 6 | 3 | 3
ng*hr/mL | 220.1116 (47.966) | 240.1012 (38.261) | 322.9544 (51.178) | 276.9650 (74.314) | 1590.2451 (38.770) | 2690.2403 (45.633)

16. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From 0 to Infinity for TAK-228 on Cycle 1 Day 1
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 3 | 3
ng*hr/mL | 143.6467 (51.931) | 204.3414 (36.134) | 320.7879 (44.795) | 192.1438 (41.892) | 1636.7944 (49.906) | 2010.7676 (53.638)

17. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The CBR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD). BOR was defined as the best response recorded after the first dose of study drug until subsequent therapy. As per Response Evaluation Criteria Solid Tumors (RECIST) version 1.1 guidelines, CR was defined as disappearance of all target lesions and non-target lesions, and normalization of tumor marker level. PR was defined as >= 30% decrease in the sum of the longest diameter (LD) of target lesions, no progression in non-target lesion, and no new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression (PD). PD was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline Up to 1 Year 7 Months
Population: The safety set includes all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 3 | 3
Percentage of participants | 33 | 50 | 57 | 33 | 67 | 67

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug and no more than 30 days after the last dose of study drug (up to Cycle 12 Day 58)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/7 | 0/6 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 3/7 | 1/6 | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg (N=3) | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg (N=6) | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg (N=7) | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg (N=6) | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg (N=3) | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg (N=3)
Genital Herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation, Daily Dosing Arm: TAK-228 2 mg (N=3) | Dose Escalation, Daily Dosing Arm: TAK-228 3 mg (N=6) | Dose Escalation, Daily Dosing Arm: TAK-228 4 mg (N=7) | Dose Expansion, Daily Dosing Arm: TAK-228 3 mg (N=6) | Dose Escalation, Weekly Dosing Arm: TAK-228 20 mg (N=3) | Dose Escalation, Weekly Dosing Arm: TAK-228 30 mg (N=3)
Stomatitis (Gastrointestinal disorders) | 0 | 5 | 4 | 5 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rash erythmatous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 3 | 3 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1 | 2 | 2 | 1
Platelet count decreased (Investigations) | 0 | 1 | 2 | 3 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 2 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 0 | 2 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 3 | 0 | 0
Gamma-glutamyltransferase increases (Investigations) | 0 | 0 | 0 | 2 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 4 | 4 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 3 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 3 | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 2 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Cystitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 4 | 2 | 3 | 3
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT03370302/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03370302/SAP_001.pdf